CLINICAL TRIAL: NCT05347953
Title: Gravitational Arrhythmogenesis Can the Often-heard Symptom of Body Position Dependent Palpitations be Proven
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Maarten van den Broek, JLPM van den Broek, MD, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL 81272.100.22
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Complexes, Premature; Atrial Fibrillation
Keywords: Body position
MeSH Terms: conditions — Cardiac Complexes, Premature; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm: Patients with self-reported symptoms of positional dependent palpitations
  Interventions: Device: Single night downgraded home polygraphy

INTERVENTIONS:
Device: Single night downgraded home polygraphy — All patients will be outfitted with the ambulatory downgraded polygraphy device (Nox A1, Nox Medical Global, Reykjavik) for 24 hour monitoring. The data exported by the polygraphy device is in European Data Format and will be filtered and annotated using custom MATLAB-software.

SUMMARY:
This study aims to assess the relationship between body position and the occurrence of either atrial or ventricular premature beats and more complex arrhythmia

DETAILED DESCRIPTION:
Rationale: Palpitations in a certain body position is an often-heard symptom, although there is currently no direct evidence that links body position with arrhythmia. The hypothesis is that arrhythmia is more prevalent in the specific body position that the patient reports to be arrhythmogenic.

Objective: The objective of this study is to assess the relationship between body position and the occurrence of either atrial or ventricular premature beats and more complex arrhythmia (AT, atrial fibrillation (AF), VT) in a population that have a self-reported preferential body position for symptoms.

Study design: Single cohort study. Subjects are recruited from the outpatient clinic. First, they will fill in a short questionnaire regarding their symptoms; second, they will be outfitted with a downgraded polygraphy device, that only monitors body position, and single and/or multi lead ECG for 24 hours. The acquired data will be analyzed at the Catharina Hospital and the Eindhoven University of Technology.

Study population: Outpatients with palpitations and a self-reported higher prevalence in a certain body position that have an indication to undergo Holter monitoring, independent of any previous diagnosis.

Main study parameters/endpoints: The frequency of ectopic beats or onset of complex arrhythmia (n per minute) in the body position that the patient has reported as arrhythmogenic, compared to arrhythmia rate in the other body positions, corrected for time spent per body position.

ELIGIBILITY:
Inclusion Criteria:

* Palpitations, spontaneously described to occur either predominantly or solely in a certain body position (upright, prone, supine, left or right lateral decubital position).
* Ability to provide informed consent

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in outpatients that present with palpitations and a spontaneous self-reported higher prevalence in a certain body position.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia per body position | 1 night recording
  The frequency of ectopic beats or onset of complex arrhythmia (n per minute) in the body position that the patient has reported as arrhythmogenic, compared to arrhythmia rate in the other body positions, corrected for time spent per body position.

CONTACTS AND LOCATIONS:
Overall Officials: JLPM van den Broek, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be available upon reasonable request by non-commercial fellow researchers
Supporting Information: Study Protocol, SAP
Time Frame: 1-20 years after publication of study
Access Criteria: non-commercial